CLINICAL TRIAL: NCT05436392
Title: DROP-Benzo (De-adopting Routine Preoperative Benzodiazepines for Older Surgical Patients): a Randomized Trial of Behavioral Strategies to Reduce Unnecessary Midazolam Administration to Older Surgical Patients
Brief Title: De-adopting Routine Preoperative Benzodiazepines for Older Surgical Patients
Acronym: DROP-Benzo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: US Anesthesia Partners (Unknown); Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Mark Neuman, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 850809
Record Dates: First submitted 2022-06-02; First posted 2022-06-29 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Surgery; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention)
- Peer Comparison Feedback (Experimental)
  Interventions: Behavioral: Peer Comparison Feedback
- Patient Informational Letter (Experimental)
  Interventions: Behavioral: Patient Informational Letter
- Peer Comparison Feedback plus Patient Informational Letter (Experimental)
  Interventions: Behavioral: Peer Comparison Feedback; Behavioral: Patient Informational Letter

INTERVENTIONS:
Behavioral: Peer Comparison Feedback — USAP anesthesia providers will receive monthly alerts via USAP's smartphone-based practice management application, text message, or email presenting individual-level data on their benzodiazepine administration patterns versus other USAP providers, using data from the USAP clinical and quality data warehouse.
  Arms: Peer Comparison Feedback; Peer Comparison Feedback plus Patient Informational Letter
Behavioral: Patient Informational Letter — Breif informational letters will be distributed to eligible patients within the 2 weeks prior to surgery. Letters will be produced on USAP letterhead and signed by the USAP Chief Quality Officer. Letter text will state USAP's commitment to brain health and avoiding potentially unnecessary medications for patients undergoing surgery. It will also include a statement encouraging patients to discuss anesthesia plans with their clinicians at the time of surgery to aid tailoring of care to individual needs. Letters will be distributed directly to patients via text link, email, or hard copy as a component of standard pre-operative instructional communications and other educational and patient outreach materials related to clinical care.
  Arms: Patient Informational Letter; Peer Comparison Feedback plus Patient Informational Letter

SUMMARY:
Over 21 million surgical procedures take place among adults aged 65 and older in the US each year, and most older surgical patients in the US now receive benzodiazepines (e.g., midazolam, lorazepam) during anesthesia care. This occurs despite recommendations to avoid these medications in older patients due to associated medical risks and lack of demonstrated benefit. In other words, routine benzodiazepine administration to older surgical patients is likely to represent low-value care that is a suitable target for de-adoption. In this study, we will evaluate a United States Anesthesia Partners (USAP, Dallas, TX) quality improvement initiative using peer comparison feedback to clinicians and/or mailed informational letters to patients as strategies to encourage physician de-adoption of routine preoperative benzodiazepine administration to older surgical patients. In partnership with USAP, this study will be conducted using randomization to evaluate its effect.

ELIGIBILITY:
Inclusion Criteria:

* All anesthesia clinicians employed by USAP will be included in the evaluation. Patients will be included if they are at least aged 65 and undergo an elective (scheduled) surgical or endoscopic procedure under general anesthesia.

Exclusion Criteria:

* Patients will be excluded if they are unscheduled (urgent/emergent) cases due to inability to reliably deliver study interventions to this group; if they did not receive general anesthesia; or if they received a nerve block procedure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 517611 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Benzodiazepine administration rate | Intraoperative period
  The primary outcome measure is the change in the rate of benzodiazepine administration among eligible surgical cases.

SECONDARY OUTCOMES:
Patient satisfaction | Up to 30 days after surgery
  Change in patient satisfaction with care, as measured by Anesthesiologist Patient Satisfaction Questionnaire Composite Satisfaction Score, Version 2 (APSQ2).

OTHER OUTCOMES:
Hospital length of stay | Length of stay will be evaluated at approximately 30 days after surgery
  Time from surgery to hospital discharge in days
Postoperative pulmonary complications | Up to 30 days after surgery
  Postoperative pulmonary complications as identified by ICD-10 codes for patients undergoing hospitalization after surgery
Postoperative Delirium | Up to 30 days after surgery
  Postoperative delirium as identified by ICD-10 codes for patients undergoing hospitalization after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Neuman, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- US Anesthesia Partners, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neuman MD, Feng R, Shukla AS, Han X, Horan AD, Whatley K, Schapira MM, Marcantonio ER, Dutton RP. Strategies to Limit Benzodiazepine Use in Anesthesia for Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2442207. doi: 10.1001/jamanetworkopen.2024.42207. PMID 39480422